CLINICAL TRIAL: NCT07133555
Title: Expanding Safe Spaces 4 Sexual Health, a Mobile Van HIV/STI Testing and Care Linkage Strategy, for MSM in Online Spaces
Brief Title: Safe Spaces 4 Sexual Health
Acronym: SS4SH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00442069
Record Dates: First submitted 2025-08-12; First posted 2025-08-21 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: HIV Counseling and Testing; HIV Risk Behavior; HIV Prevention
Keywords: geosocial networking application; peer health coach; peer health navigator; hiv mobile testing; black msm; online spaces; linkage to HIV treatment; linkage to HIV prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group receiving peer health navigation follow-up (Experimental): Participants randomly assigned to Arm A will receive a navigation/care linkage needs assessment followed by peer navigation once weekly after discussing their test results with the navigator to support their linkage to PrEP or HIV care over a six-week period. Navigators will complete the following care linkage steps: 1) assess interest in linkage, 2) identify preferred clinic for care linkage, and 3) assist with scheduling initial PrEP/HIV provider appointment. Additionally, the investigators will use the qualitative data collected from in-depth interviews (IRB00375934) of Black MSM and key informant interviews of care linkage stakeholders on barriers and facilitators to HIV prevention and care linkage strategies to inform the peer navigation that Arm A receives.
  Interventions: Other: Healthcare counseling service
- Control group receiving standard of care referral (No Intervention): Participants randomly assigned to Arm B will go through the standard of care referral process to a local community site providing PrEP or HIV care after discussing their test results with a navigator. During this discussion with a navigator, participants will receive information about the PrEP/HIV care sites where the participants can go for services. Six weeks following this initial follow-up, participants will meet virtually with the navigator to complete a PrEP/care linkage status assessment to determine if the participants attended the initial PrEP/HIV provider appointment.

INTERVENTIONS:
Other: Healthcare counseling service — Using peer health navigators to support linkage to HIV prevention and treatment resources among Black MSM in online spaces following mobile testing.
  Arms: Intervention group receiving peer health navigation follow-up

SUMMARY:
In an earlier study, the study team carried out an HIV/Sexually transmitted infection (STI) testing approach which found men who have sex with men (MSM) at-risk of getting or spreading HIV in online spaces and linked them to testing services on a mobile van. The goal of this present study is to add on to this approach by connecting participants (MSM aged 18-49 residing in the Baltimore area) with a peer health navigator to support them with getting pre-exposure prophylaxis (PrEP) or HIV care services after testing. Researchers will compare using a peer health navigator approach to using a referrals-only approach to get PrEP or HIV care services. Participants will be assigned to either Arm A (group that receives peer health navigator help) or Arm B (group that gets referred) to get PrEP or HIV care.

DETAILED DESCRIPTION:
In the SS4SH pilot study, utilizing a data-driven approach in partnership with the local health department, the investigators analyzed local public health surveillance data to identify online sex partner meeting spaces frequently reported by (majority Black) MSM newly diagnosed with HIV and/or syphilis. The identified online spaces were used to advertise mobile van HIV/STI testing for MSM > 18 years of age and less than 49 years of age over a 14-month period. The strategy and advertisements were informed by a community advisory board (CAB) of MSM hosted at a local Lesbian, Gay, Bisexual, Transgender, and Queer (LGBTQ) community-based organization to ensure local relevance, acceptability and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-49 years of age
* Ability to read and speak English
* Baltimore area resident
* Report sex with a male in the past 12 months

Exclusion Criteria:

* not male-self identified individual

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male self-identified individuals are eligible to participate.
Enrollment: 100 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of adding care linkage assessed by retention rate | 6 weeks
  Feasibility of adding care linkage will be measured based on the retention rate during follow-up period of Arm A participants in need of PrEP/HIV care linkage. Retention rate of 75% will be used as a feasibility threshold. Linkage is defined as completing a PrEP/HIV care related medical visit within 30 days of enrollment.
Acceptability as assessed by participant satisfaction | 6 weeks
  A satisfaction rate of 75% or greater will be used as the acceptability threshold.
Acceptability as assessed by number of participants with intent to repeat use of SS4SH | 6 weeks
  Acceptability will be measured as intention for repeat use of SS4SH testing/care linkage modality.
Effectiveness as assessed by the number of Black MSM linked to HIV/PrEP | 30 days
  Preliminary data on effectiveness will be assessed by number of Black MSM linked to HIV care and PrEP within 30 days of enrollment. Linkage is defined as completing a PrEP/HIV care related medical visit.
Effectiveness as assessed by number of Black MSM lost to followup | 30 days
  Preliminary data on Effectiveness assessed by number of Black MSM lost to follow up. Linkage is defined as completing a PrEP/HIV care related medical visit.

SECONDARY OUTCOMES:
Reach/awareness of the geotargeted advertisement campaign assessed by cost per 1,000 impressions (CPM) | 12 weeks
  Defined by impressions, cost per 1,000 impressions (CPM)
Website traffic of the geotargeted advertisement campaign assessed by cost per click (CPC) | 12 weeks
  Defined by clicks, cost per click (CPC)
Cost per action conversion rate of the geotargeted advertisement campaign | 12 weeks
  Actions will include website actions (view schedule, scheduling appointments) and van actions (HIV/STI testing)

CONTACTS AND LOCATIONS:
Overall Officials: Errol L Fields, MD, PhD, MPH, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fields EL, Thornton N, Huettner S, Schumacher C, Barrow G, Greenbaum A, Jennings JM. Safe Spaces 4 Sexual Health: A Status-Neutral, Mobile Van, HIV/STI Testing Intervention Using Online Outreach to Reach MSM at High Risk for HIV Acquisition or Transmission. J Acquir Immune Defic Syndr. 2022 Jul 1;90(S1):S84-S89. doi: 10.1097/QAI.0000000000002968. PMID 35703759
- [Background] Rosenberg ES, Millett GA, Sullivan PS, Del Rio C, Curran JW. Understanding the HIV disparities between black and white men who have sex with men in the USA using the HIV care continuum: a modeling study. Lancet HIV. 2014 Dec;1(3):e112-e118. doi: 10.1016/S2352-3018(14)00011-3. PMID 25530987
- [Background] Oster AM, Wiegand RE, Sionean C, Miles IJ, Thomas PE, Melendez-Morales L, Le BC, Millett GA. Understanding disparities in HIV infection between black and white MSM in the United States. AIDS. 2011 May 15;25(8):1103-12. doi: 10.1097/QAD.0b013e3283471efa. PMID 21505305